CLINICAL TRIAL: NCT06108570
Title: Evaluation of the Efficacy and Tolerance of TOPIALYSE Baume Protect+ Vs Neutral Product on Patients Suffering from Atopic Dermatitis
Brief Title: Evaluation of the Efficacy of TOPIALYSE Baume Protect+ on Atopic Dermatis
Acronym: TOPIAbis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SVR Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOPIAbis-2022; B4032023000074 (Other: Belgium)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison
Masking Description: The randomisation will be done on the side of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study methodology (Other): This is an intra-individual comparison study.
  Interventions: Other: Cosmetic Product TOPIALYSE Baume Protect+

INTERVENTIONS:
Other: Cosmetic Product TOPIALYSE Baume Protect+ — One or two application.s of TOPIALYSE Baume Protect+ daily on one side for 28±3 days and the Neutral Product daily on the other side for 28±3 days. The side will be decided before by randomisation.
  Other Names: Cosmetic product Neutral Product

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of a SVR care product.

As we know, atopic dermatitis is a vicious circle that must be broken, but certain aggravating factors are added to this circle. There is a lot of talk about pollution but, more recently, studies have been carried out on the worsening role of dust mites on atopic skin.

TOPIALYSE Baume Protect+ is a care product that is lipid-replenishing, repairing and protective: a triple reinforced action for 48 hours: anti-scratching, anti-irritation, and external anti-aggression. It is also intended for the whole family from birth for dry skin with an atopic tendency (with atopic eczema).

The main objective of this study is to evaluate the efficacy of the cosmetic product SVR TOPIALYSE Baume Protect+ versus Neutral Product on patients with mild atopic dermatitis, after 4 weeks of use with evaluation of the evolution mEASI (modified Eczema Area and Severity Index)

DETAILED DESCRIPTION:
1. RATIONALE : The purpose of this study is to evaluate the efficacy and tolerability of a SVR care product.

As we know, atopic dermatitis is a vicious circle that must be broken, but certain aggravating factors are added to this circle. There is a lot of talk about pollution but, more recently, studies have been carried out on the worsening role of dust mites on atopic skin.

The new SVR product, TOPIALYSE Baume Protect+ will therefore be based on it.

TOPIALYSE Baume Protect+ is a care product that is lipid-replenishing, repairing and protective: a triple reinforced action for 48 hours: anti-scratching, anti-irritation, and external anti-aggression. It is also intended for the whole family from birth for dry skin with an atopic tendency (with atopic eczema).

2 STUDY OBJECTIVES 2.1 PRIMARY OBJECTIVE: The main objective of this study is to evaluate the efficacy of the cosmetic product SVR TOPIALYSE Baume Protect+ versus Neutral Product on patients with mild atopic dermatitis, after 4 weeks of use with evaluation of the evolution mEASI (modified Eczema Area and Severity index ).

2.2 SECONDARY OBJECTIVE:

- To assess the tolerance of TOPIALYSE Baume Protect+ versus Neutral Product by a scale of 0 to 5, (0 corresponding to no reaction and 5 to severe) after 4 weeks of application.

* To assess the product's efficacy in improving children's quality of life using the IDQOL questionnaire (Infant's Dermatitis Quality of Life index ).
* To assess the efficacy of the product on the reduction of pruritus using the Visual Analog Scale (VAS).
* Taking of close-up photographs of the lesions / anonymized when the patients or their parent(s) have given their consent.
* Analysis of the subjects' answers to a subjective product evaluation questionnaire.

  3.STUDY METHODOLOGY This is a multicentric, randomized, intra-individual and double-blind study. It is an interventional study with minimal risks (Category 2).

3.1 EVALUATION CRITERIA 3.1.1 Primary criteria • Evaluation of the efficacy of the product by reducing the symptoms associated with mild atopic dermatitis with evaluation of the evolution of the mEASI (modified Eczema Area and Severity index).

3.1.2 Secondary criteria

* Assessment of the tolerance of TOPIALYSE Baume Protect+ versus Neutral Product on a scale of 0 to 5, (0 corresponding to no reaction and 5 to severe) after 4 weeks of application.
* Assessment of the product's efficacy in improving children's quality of life using the IDQOL questionnaire (Infant's Dermatitis Quality of Life index).
* Evaluation of the efficacy of the product on the reduction of pruritus using the Visual Analog Scale (VAS).
* Taking of close-up photographs of the lesions / anonymized when the patients or their parent(s) have given their consent.
* Analysis of the subjects' answers to a subjective product evaluation questionnaire.
* General safety: General Adverse Events will be reported descriptively on an on-going basis.

3.2 EVALUATION METHODS

3.2.1 Modified Eczema Area and Severity Index At D0 and D28±3, the dermatologist calculates the mEASI over the entire body. A. First, the investigator selects the affected areas. B. For each zone, the investigator assesses the severity of the 4 signs of atopic dermatitis (erythema, oedema/papulation, excoriation, lichenification) from 0 to 3 on the selected area.

C. For each zone, the investigator assesses the extent of atopic dermatitis in that area.

D. Then the investigator will obtain the mEASI score of each area after applying the multiplying factor. The multiplying factor may be different if the patient is less than 8 years old.

3.2.2 IDQOL At D0 and D28±3, the dermatologist calculates the SCORE IDQOL using the Quality-of-Life Questionnaire on Early Childhood Eczema completed by the parents.

To obtain the IDQOL score, the investigator adds up the scores given for each response with a maximum of 30 and a minimum of 0. The higher the score, the greater the impact on quality of life. The severity of eczema is scored separately and can be correlated with the IDQOL score.

3.2.3 Pruritus assessment Pruritus will be assessed using the visual analogue scale VAS at Day 0 before product application and at Day 28±3.

3.2.4 Subjective evaluation questionnaire A subjective evaluation questionnaire is completed by subjects at D28±3 to subjectively assess the efficacy and acceptability of the product studied.

3.2.5 Standardized photographs Standardized photographs of the affected areas (body and/or face) if authorized and desired will be performed at D0 and D28±3

4.Duration of treatment The tested products will be applied for twenty-eight to thirty-one days consecutively.

5.Dose For the test products an amount of about 2mg/cm² on a whole child body test area (0,46m² (1-year-old babies) to 1,85m² (adolescents) area [25]) will be applied once a day or twice a day. The subject will be shown the amount of product to be applied.

6 INVESTIGATIONAL PLAN 6.1 STUDY DESIGN This is a multicentric, randomized, intra-individual and double-blind study. It is an interventional study with minimal risks (Category 2).

The study will be performed in sixty children with mild atopic dermatitis, seventy-two (72) will be pre-screened if we consider a risk of approximately 20% drop-out. The screening of the subjects will be performed at the investigator's medical office within three months prior to the first study visit (at Day 0) and to allow verification of the subject compatibility with the inclusion and exclusion criteria. During the screening visit a physical examination and vital sign measurement will be performed.

6.1.1 Study location The study will be performed in five Investigation centers.

6.1.2 Study duration The study participation for each subject will last up to 1 month (28±3 days of clinical participation).

6.2 STUDY PROCEDURES 6.2.1 Screening visit: The screening visit will be performed within three months of the day before Day 0. The following procedures may be carried on several days if needed.

* Subject information and presentation of the informed consent form,
* Inclusion/ exclusion criteria checking.

6.2.2 Visit 1 Baseline: Day 0

The subject will have to come to the investigator site for:

* Signing the consent form
* Verification of inclusion and non-inclusion criteria
* Clinical examination / Medical history
* Randomization
* Complete source file and CRF
* mEASI clinical scoring
* IDQOL questionnaire
* Assessment of pruritus with the VAS
* Taking of standardized photographs if applicable
* Distribution of products in relation to randomization
* Weigh study products and record in the source file and CRF
* Distribution of logbook and patient card
* First application of products in office (left/right)
* Schedule next appointment for D28-D31.

Between this visit and the next:

* Use of the products
* Daily filling of the logbook.

6.2.3 Visit 2, Follow-up and the end of the study: Day 28±3

* Verification of the patient logbook
* Follow-up of adverse events, intolerance and associated treatments
* Fill in the source file and the CRF
* mEASI clinical scoring
* IDQOL questionnaire
* Evaluation of pruritus with the VAS scale
* Taking of standardized photographs if applicable
* Subjective evaluation questionnaire
* Collection of follow-up booklets
* Collection of study products
* Weigh the products and record in the source file and CRF
* End of study. After this visit, the patients will stop using the TOPIALYSE Baume Protect+ emollient and the neutral product.

  8 STATISTICAL METHODS 8.1 BASELINE CHARACTERISTICS Continuous demographic variables (e.g. age, weight, and height) will be summarized, using mean, standard deviation, minimum, maximum and number of available observations.

Qualitative demographic characteristics will be summarized by counts and percent. Other subject characteristics (anomalies in physical examination, prior medication, inclusion / exclusion checklist) will be listed only.

8.2 PRIMARY CRITERION

• Evaluation of the efficacy of the product by reducing the symptoms associated with mild atopic dermatitis with evaluation of the evolution of the mEASI (modified Eczema Area and Severity Index)

8.3 SECONDARY CRITERIA

* Evaluation of the tolerance of TOPIALYSE Baume Protect+ versus Neutral Product by a scale of 0 to 5, (0 corresponding to no reaction and 5 to severe) after 4 weeks of application.
* Evaluation of the product's efficacy in improving children's quality of life using the IDQOL questionnaire (Infant's Dermatitis Quality Of Life index).
* Evaluation of the efficacy of the product on the reduction of pruritus using the Visual Analog Scale (VAS).
* Taking of close-up photographs of the lesions / anonymized when the patients or their parent(s) have given their consent.
* Analysis of the subjects' answers to a subjective product evaluation?questionnaire.
* General safety: General Adverse Events will be reported descriptively on an on-going basis.

8.4 STATISTICAL ANALYSES Descriptive statistics (N, mean, standard error, min, max,) will be calculated by test product for each parameter.

Prior to any statistical analysis, the normality of each variable will be tested using the Shapiro Wilks test of normality.

Statistical Tests For each normal variable, comparisons will be performed using a t-test for paired data.

For each non normal variable, comparison will be performed using a Wilcoxon rank sum test.

8.5 NUMBER OF SUBJECTS CALCULATION The expected benefit is an improvement in the severity of atopic dermatitis with a decrease in EASI / mEASI.

A literature review shows that for a mean baseline EASI of 4.49, patients with mild to moderate atopic dermatitis treated with a class 1 topical medical device enriched with antioxidants twice daily for 28 days [26] showed a decrease of this score of 3.41 (standard deviation of the baseline population = 3.87). We expect similar results given the compositions of the medical device and the tested product, as well as a slighter effect with the placebo (decrease of about 0.5 with the placebo). These different parameters define a Cohen effect size of d=0.75, i.e., a strong effect. A calculation of the number of subjects shows that with an α level of 0.05 (one-sided) and a power of 80%, we obtain a total number of subjects of 46. A minimum of 23 patients per group would therefore be needed according to this scheme.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer aged between 3 months and 18 years
2. Female or male volunteer
3. Volunteer with an atopic background and localized and symmetrical right/left signs of mild atopic dermatitis on the face and/or body: On the whole body: 0.1 < EASI < 7 [2] or

   Localized - mEASI (cf. Appendix n°1):
   * On the arms: 0.02 < mEASI < 1.4
   * On the legs: 0.04 < mEASI < 2.8 (0.03 < mEASI < 2.1 for children under 8 years old)
   * On the trunk: 0.03 < mEASI < 2.1
   * On the head/neck: 0.01 < mEASI < 0.7 (0.02 < mEASI < 1.4 for children under 8 years old)
4. Volunteer agreeing not to use any other skincare product on the face or body for the duration of the study, except for study products,
5. Volunteer agreeing not to perform any corticosteroid or immunosuppressive treatment, per os or topical for the duration of the study,
6. Volunteer whose parent(s) or legal guardian(s) have given written consent to participate in the study,
7. Volunteer related to the social security of a parent or legal guardian in accordance with the French law on interventional research

Exclusion Criteria:

1. Volunteer with a history of allergy or hypersensitivity reaction to a cosmetic or any of the constituents of the test products.
2. Volunteer who received topical corticosteroid or immunosuppressive treatments during the week prior to study entry and during the study.
3. Volunteer who received oral corticosteroids during the month prior to study entry.
4. Presence of dermatosis, skin pathology or systemic disease that, in the opinion of the investigator, may interfere with the evaluation of the study parameters.
5. Existence of a systemic or local treatment which, in the opinion of the investigator, may interfere with the evaluation of the parameters studied.
6. Volunteer participating in another study or being in an exclusion period from a previous study.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of the evolution of the symptoms associated with mild atopic dermatitis by the mEASI score | DAY 0 and DAY 28±3
  At D0 and D28±3, the dermatologist calculates the mEASI (modified Eczema Area and Severity Index) over the entire body, for that he have to select the affected area ( head and neck, upper extremities, trunk, lower extremities). For each zone, the investigator assesses the severity of the 4 signs of atopic dermatitis (erythema, oedema/papulation, excoriation, lichenification) from 0 ( none) to 3 (severe) on the selected area, he assesse the extent of atopic dermatitis in that area from 0 (none) to 6 (100% area of the body).

SECONDARY OUTCOMES:
Evaluation of the tolerance of TOPIALYSE Baume Protect+ versus Neutral Product. | DAY 28±3
  Evaluation of the tolerance of TOPIALYSE Baume Protect+ versus Neutral Product by a scale of 0 to 5, (0 corresponding to no reaction and 5 to severe) after 4 weeks of application.
Evaluation of children's quality of life by IDQOL | DAY 0 and DAY 28±3
  Assessing the product's impact on enhancing the quality of life for children using the IDQOL (Infant's Dermatitis Quality Of Life index )questionnaire. To obtain the IDQOL score, the investigator adds up the scores given for each response with a maximum of 30 and a minimum of 0. The higher the score, the greater the impact on quality of life
Evaluation of pruritus by VAS | DAY 0 and DAY 28±3
  Evaluation of the efficacy of the product on the reduction of pruritus using the Visual Analog Scale (VAS), on a scale from "no itch" (left) to "most itchy unbearable" (right), at DAY 28±3 versus DAY 0 before product application.
Analysis of the subject's answers to a subjective product evaluation questionnaire | DAY 0 and DAY 28±3
  A subjective evaluation questionnaire is completed by subjects to subjectively assess the efficacy and acceptability of the product studied by responding with (Quite All right), (All right), (Not quite All right), (Not All right), at DAY 28±3 versus DAY 0
General safety: General Adverse Events will be reported descriptively on an on-going basis | DAY 0 and DAY 28±3
  General safety: General Adverse Events will be reported descriptively on an on-going basis, at DAY 0 versus DAY 28±3. (Follow-up of the number of Adverse Events especially those linked with the products).

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hopital Universitaire Des Enfants Reine Fabiola, Brussels
  - Grand Hopital de Charleroi, Charleroi

IPD SHARING:
Plan to Share IPD: No